CLINICAL TRIAL: NCT04042701
Title: A Phase 1b, Multicenter, Two-Part, Open-Label Study of Trastuzumab Deruxtecan (DS-8201a), An Anti-Human Epidermal Growth Factor Receptor-2 (HER2)-Antibody Drug Conjugate (ADC), In Combination With Pembrolizumab, An Anti-PD-1 Antibody, For Subjects With Locally Advanced/Metastatic Breast Or Non-Small Cell Lung Cancer (NSCLC)
Brief Title: DS8201a and Pembrolizumab in Participants With Locally Advanced/Metastatic Breast or Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-U106; 2018-002489-38 (EudraCT Number); KEYNOTE-797 (Other: Merck Sharp & Dohme Corp); MK-3475-797 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Non-small Cell Lung Carcinoma
Keywords: Human epidermal receptor 2 positive; Human epidermal receptor 2; Non-small Cell Lung Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — trastuzumab deruxtecan; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase 1b, open-label, 2-part, multicenter, non-randomized, multiple-dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Part 1 (Dose Escalation) (Experimental): HER2-positive breast cancer, HER2-low expressing breast cancer, HER2-expressing NSCLC, and HER2-mutant NSCLC participants who received escalating doses of DS8201a (initial dose 3.2 mg/kg Q3W) and pembrolizumab 200 mg.
  Interventions: Drug: Trastuzumab deruxtecan (DS-8201a); Drug: Pembrolizumab
- HER2-positive breast cancer (Part 2 Dose Expansion) (Experimental): HER2-positive breast cancer participants with prior ado-trastuzumab emtansine (T-DM1) with disease progression and who received DS8201a at the RDE in combination with pembrolizumab 200 mg.
  Interventions: Drug: Trastuzumab deruxtecan (DS-8201a); Drug: Pembrolizumab
- HER2-low breast cancer (Part 2 Dose Expansion) (Experimental): HER2 low breast cancer participants with prior failed standard treatments who received DS8201a at the RDE in combination with pembrolizumab 200 mg.
  Interventions: Drug: Trastuzumab deruxtecan (DS-8201a); Drug: Pembrolizumab
- HER2-expressing NSCLC (Part 2 Dose Expansion) (Experimental): HER2-expressing NSCLC participants who had not received any prior treatment with anti-PD-1, anti-PD-L1, or HER2 agents and received DS8201a at the RDE in combination with pembrolizumab 200 mg.
  Interventions: Drug: Trastuzumab deruxtecan (DS-8201a); Drug: Pembrolizumab
- HER2-mutant NSCLC (Part 2 Dose Expansion) (Experimental): HER2-mutant NSCLC participants who had not received any prior treatment with anti-PD-1, anti-PD-L1, or HER2 agents and received DS8201a at the RDE in combination with pembrolizumab 200 mg.
  Interventions: Drug: Trastuzumab deruxtecan (DS-8201a); Drug: Pembrolizumab

INTERVENTIONS:
Drug: Trastuzumab deruxtecan (DS-8201a) — Part 1: Two dose levels of DS-8201a (3.2 mg/kg Q3W and 5.4 mg/kg Q3W via intravenous (IV) infusion will be administered for the dose escalation part of the study in combination with pembrolizumab.
  Part 2: Once Part 1 of the study is complete and a RDE for DS-8201a has been established, Part 2 will begin. All participants will receive DS-8201a at the RDE in combination with pembrolizumab.
  Arms: HER2-expressing NSCLC (Part 2 Dose Expansion); HER2-low breast cancer (Part 2 Dose Expansion); HER2-mutant NSCLC (Part 2 Dose Expansion); HER2-positive breast cancer (Part 2 Dose Expansion)
Drug: Trastuzumab deruxtecan (DS-8201a) — Part 1: Two dose levels of DS-8201a (3.2 mg/kg Q3W and 5.4 mg/kg Q3W via intravenous (IV) infusion will be administered for the dose escalation part of the study in combination with pembrolizumab.
  Part 2: Once Part 1 of the study is complete and a RDE for DS-8201a has been established, Part 2 will begin.
  Arms: Part 1 (Dose Escalation)
Drug: Pembrolizumab — All participants will receive pembrolizumab (200 mg Q3W) via intravenous (IV) infusion prior to DS-8201a in Parts 1 and 2 of the study.
  Other Names: KEYTRUDA®

SUMMARY:
This two-part study will include a dose escalation part to determine the recommended dose for expansion of DS8201a and pembrolizumab and a dose expansion part to evaluate efficacy, safety, and tolerability of the combination.

DETAILED DESCRIPTION:
This phase 1b, open-label, 2-part, multicenter, non-randomized, multiple-dose study will evaluate DS-8201a in combination with pembrolizumab in participants with advanced/metastatic breast cancer or non-small cell lung cancer (NSCLC).

In the dose escalation part of the study, escalating doses of DS-8201a in combination with pembrolizumab will be assessed. DS-8201a and pembrolizumab 200 mg will be administered on Day 1 of every 21-day cycle. The initial dose administered for DS8201a will be 3.2 mg/kg Q3W. Escalation to the next dose (5.4 mg/kg Q3W) will be based on acceptable safety signals based on the earlier dose cohort.

Upon completion of dose escalation with the recommended dose of escalation (RDE) established, the dose expansion part of the study will begin. The dose expansion part will include 4 cohorts: Human epidermal growth factor receptor 2 (HER2+) breast cancer participants with prior ado-trastuzumab emtansine (T-DM1), HER2 low breast cancer participants with prior failed standard treatments, HER2-expressing NSCLC participants who have not received any prior treatment with anti-PD-1, anti-PD-L1, or HER2 agents, and HER2-mutant NSCLC participants who have not received any prior treatment with anti-PD-1, anti-PD-L1, or HER2 agents.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adults ≥18 years
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 to 1
* Pathologically documented HER2-expressing locally advanced/metastatic breast cancer, and HER2-expressing or HER2-mutant locally advanced/metastatic NSCLC
* Willing to provide a tumor biopsy during screening and during treatment
* Have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as assessed by the Investigator
* Adequate cardiac function, as defined by left ventricular ejection fraction (LVEF) ≥50% within 28 days before enrollment.
* Adequate organ function
* Adequate treatment washout period before enrollment

Inclusion Criteria Specific to Part 1

* Participants in Part 1 should meet the additional inclusion criteria listed for 1 of the 4 cohorts in Part 2.

Inclusion Criteria Specific to Part 2

Inclusion Criteria for Cohort 1

* Pathologically documented, locally advanced/metastatic breast cancer that has centrally determined HER2-positive expression as per American Society of Clinical Oncology-College of American Pathologists (ASCO-CAP) Guidelines
* Received prior trastuzumab emtansine (T-DM1) therapy with documented progression

Inclusion Criteria for Cohort 2

* Pathologically documented, locally advanced/metastatic breast cancer that has centrally determined HER2-low expression (immunohistochemistry [IHC] 1+ or IHC 2+/in situ hybridization [ISH-])
* Participants must have exhausted treatments that can confer any clinically meaningful benefit (eg, other therapies such as hormonal therapy for participants who are hormone receptor positive)

Inclusion Criteria for Cohort 3

* Pathologically documented, locally advanced/metastatic NSCLC that has centrally or locally determined HER2-expression (IHC 1+, 2+, or 3+)
* Participants who have known epidermal growth factor receptor (EGFR) mutation, anaplastic lymphoma kinase (ALK), BRAF V600E mutation, or ROS1 fusion should have disease progression after treatment with at least one genomically-targeted therapy for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment

Inclusion Criteria for Cohort 4

* Pathologically documented, locally advanced/metastatic HER2-mutant NSCLC
* Participants who have known EGFR mutation, ALK, BRAF V600E mutation, or ROS1 fusion should have disease progression after treatment with at least one genomically-targeted therapy for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment

Exclusion Criteria:

* Prior treatment with pembrolizumab or DS-8201a
* Medical history of myocardial infarction (MI) within 6 months before enrollment, symptomatic congestive heart failure (New York Heart Association Class II to IV). Participants with troponin levels above the upper limit of normal at Screening (as defined by the manufacturer), and without any MI-related symptoms, should have a cardiologic consultation before enrollment to rule out MI
* Corrected QT interval (QTc) prolongation to >470 ms (females) or >450 ms (males)
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Spinal cord compression or clinically active central nervous system metastases
* Active, known or suspected autoimmune disease
* Condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment
* Prior therapy with an anti-PD-1 or anti-PD-L1 agent
* Prior therapy with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event (irAE)
* Prior anti-HER2 therapy is not allowed for participants with HER2 low-expressing breast cancer or participants with NSCLC (Cohorts 2, 3, or 4). Prior treatment with pan-HER tyrosine kinase inhibitor is allowed.
* Prior systemic anticancer therapy, including investigational agents within 2 to 6 weeks prior to treatment
* Unresolved toxicities from previous anticancer therapy
* Live vaccine within 30 days prior to the first dose of study drug
* Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Multiple primary malignancies within 3 years, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, other solid tumors curatively treated, or contralateral breast cancer
* History of severe hypersensitivity reactions to other monoclonal antibodies and/or any of the study drug components
* Active infection requiring systemic therapy
* Known history of human immunodeficiency virus (HIV) infection
* Active hepatitis B or C virus infection
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, or any other reason the participant is found not appropriate to participate in the opinion of the treating Investigator
* Known psychiatric or substance abuse disorders
* Prior organ transplantation, including allogeneic stem cell transplantation
* Pregnant, breastfeeding, or planning to become pregnant
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
* Uncontrolled infection requiring IV antibiotics, anti-virals, or anti-fungals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs), Part 1 | Within two 3-week cycles (6 weeks)
  Maximum Tolerated Dose (MTD) or recommended dose expansion (RDE) of DS-8201a (Part1) are based on the occurrence of DLTs.
Objective Response Rate (ORR), Confirmed by Independent Central Review, Part 2 | Within approximately 30 months

SECONDARY OUTCOMES:
Treatment-emergent adverse events | Within approximately 30 months
Pharmacokinetic Parameter Maximum Serum Concentration (Cmax) | Cycle 1, Day 1: predose and postdose, Day 8, and Day 15; Cycle 2, Day 1 predose and postdose, and Cycle 3, Day 1 (each cycle is 21 days)
  Cmax of trastuzumab deruxtecan, MAAA-118A, and total anti-HER2 antibody will be assessed.
Pharmacokinetic Parameter Area Under the Concentration-time Curve (AUC) | Cycle 1, Day 1: predose and postdose, Day 8, and Day 15; Cycle 2, Day 1 predose and postdose, and Cycle 3, Day 1 (each cycle is 21 days)
  Area under the concentration-time curve of trastuzumab deruxtecan, MAAA-118A, and total anti-HER2 antibody will be assessed.
Duration of Response (DoR) | Within approximately 30 months
Disease Control Rate (DCR) | Within approximately 30 months
Progression-Free Survival (PFS), based on Independent Central Review using RECIST v1.1 | Within approximately 30 months
Time to Response (TTR), based on Independent Central Review using RECIST v1.1 | Within approximately 30 months
Overall survival (OS) | Within approximately 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (30):
- United States (10):
  - Univ. of Cali. San Francisco Medical Center, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - Cancer Specialists of North Florida (Cbo), Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffit Cancer Center, Tampa, Florida
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Siteman Cancer Center-Washington University, St Louis, Missouri
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hope Cancer Center of East Texas, Tyler, Texas
- France (7):
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHUTimone, Marseille
  - Institut PAOLI-CALMETTES, Marsielle
  - CHU de Poitiers, Poitiers
  - Univ. du Cancer de Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif
- Spain (9):
  - Hospital Teresa Herrera (C.H.U.A.C), A Coruña
  - Inst. Oncologico Baselga Hospital Quiron, Barcelona
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hopital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital General Univ. Gregorio Marañon, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (4):
  - The Royal Marsden NHS Foundation Trust, London
  - Sarah Cannon Research Institute (SCRI), London
  - The Christie NHS Fond. Trust, Manchester
  - Royal Marsden Hosptial, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/